CLINICAL TRIAL: NCT01889004
Title: The Neural Mechanisms of Anesthesia and Human Consciousness (LOC-2013)
Brief Title: The Neural Mechanisms of Anesthesia and Human Consciousness
Acronym: LOC-2013
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Academy of Finland (Other); Hospital District of Southwestern Finland (Other)
Responsible Party: Principal Investigator, Harry Scheinin, Adjunct Professor, University of Turku
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LOC-2013; 266467 (Other Grant/Funding Number: Academy of Finland); 2013-001496-21 (EudraCT Number); KLnro 72/2013 (Registry Identifier: Finnish Medicines Agency (Fimea))
Record Dates: First submitted 2013-06-23; First posted 2013-06-28 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Consciousness, Level Altered
Keywords: Cerebral blood flow; Consciousness; Dexmedetomidine; EEG; Event related potentials; Functional magnetic resonance imaging; General anesthesia; Positron emission tomography; Propofol
MeSH Terms: conditions — Consciousness Disorders | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Experimental): Intravenous dexmedetomidine using target controlled infusion
  Interventions: Drug: Dexmedetomidine
- Propofol (Experimental): Intravenous propofol using target controlled infusion
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — Escalating concentrations until loss of responsiveness
  Other Names: Dexdor
  Arms: Dexmedetomidine
Drug: Propofol — Escalating concentrations until loss of responsiveness
  Other Names: Propofol-Lipuro
  Arms: Propofol

SUMMARY:
The explanation of consciousness poses one of the greatest challenges to science and philosophy in the 21st century. It remains unclear what consciousness is and how it emerges from brain activity. By studying anesthesia and sleep, the investigators aim to reveal what happens in the brain when consciousness is lost and when it returns. During the study, a series of Positron Emission Tomography (PET), Magnetic Resonance Imaging (MRI) and electroencephalography (EEG) studies will be carried out on healthy male subjects to reveal the neural correlates of consciousness. Consciousness of the subjects will be manipulated with normal sleep and anesthetic agents dexmedetomidine and propofol.

First, various neurophysiological tools to separate consciousness, connectedness and responsiveness during normal sleep will be tested. The most suitable methods and subjects will be selected and then tested during anesthetic-induced sedation and loss of responsiveness (LOR). The anesthetics (dexmedetomidine or propofol) will be administered as target-controlled infusions (TCI) with step-wise concentration-increments until LOR is detected. Then, TCIs are repeated in the same subjects but adjusted according to the individual drug target concentrations sufficient for LOR, and a series of PET perfusion imaging measurements will be performed to obtain the brain activity information in various states of consciousness. The same subjects will then be imaged with PET for brain activity after sleep deprivation (awake), during various sleep stages and immediately after awakening. Finally, ten dexmedetomidine subjects will be given the drug once more, and functional MRI (fMRI) data will be collected at various states of consciousness before and during verbal and nonverbal vocalizations. EEG will be continuously collected in all sessions. The depth of anesthesia will be measured using quantitative EEG and bispectral index (BIS) monitoring.

The results may lead to the discovery of new and better objective indicators of the depth of anesthesia and consciousness, and new insights into the understanding of neural mechanisms behind drug-induced loss of consciousness and ultimately the mechanisms of action of (general) anesthetics as well as consciousness itself.

DETAILED DESCRIPTION:
(not needed)

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 20-30 years
* Good general health i.e. American Society of Anesthesiologists (ASA) physical status I
* Fluent in Finnish language
* Right handedness
* Written informed consent
* Good sleep quality

Exclusion Criteria:

* Chronic medication
* History of alcohol and/or drug abuse
* Strong susceptibility for allergic reactions
* Serious nausea in connection with previous anesthesia
* Strong susceptibility for nausea
* Any use of drugs or alcohol during the 48 hours preceding anesthesia
* Use of caffeine products 10-12 hours prior the study, 24 hours before sleep studies
* Smoking
* Clinically significant previous cardiac arrhythmia / cardiac conduction impairment
* Clinically significant abnormality in prestudy laboratory tests
* Positive result in the drug screening test
* Blood donation within 90 days prior to the study
* Participation in any medical study with an experimental drug or device during the preceding 60 days
* The study subject has undergone a prior PET or SPECT study
* Any contraindication to magnetic resonance imaging (MRI)
* Hearing impairment
* Detected unsuitability based on initial electrophysiological measurements
* Detected unsuitability based on MRI scanning results
* Sleep disorder or severe sleep problem

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2014-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Regional cerebral blood flow | Several measurements during two separate days within 2 months
  Altogether 14 PET scans during two separate study days. Cerebral blood flow changes will be used as surrogates for changes in regional brain activity.

SECONDARY OUTCOMES:
EEG | Continuous data collection during five separate days within 2 months
Functional magnetic resonance imaging (fMRI) | Several measurements during one day
Event related potentials | Several time points during five separate days within 2 months

OTHER OUTCOMES:
Drug concentration in plasma | Several times points during two or three separate days within 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Harry Scheinin, MD, Principal Investigator — University of Turku
Locations (1):
- Turku PET Centre, Turku, Finland

REFERENCES:
- [Background] Langsjo JW, Alkire MT, Kaskinoro K, Hayama H, Maksimow A, Kaisti KK, Aalto S, Aantaa R, Jaaskelainen SK, Revonsuo A, Scheinin H. Returning from oblivion: imaging the neural core of consciousness. J Neurosci. 2012 Apr 4;32(14):4935-43. doi: 10.1523/JNEUROSCI.4962-11.2012. PMID 22492049
- [Derived] Valli K, Radek L, Kallionpaa RE, Scheinin A, Langsjo J, Kaisti K, Kantonen O, Korhonen J, Vahlberg T, Revonsuo A, Scheinin H. Subjective experiences during dexmedetomidine- or propofol-induced unresponsiveness and non-rapid eye movement sleep in healthy male subjects. Br J Anaesth. 2023 Aug;131(2):348-359. doi: 10.1016/j.bja.2023.04.026. Epub 2023 May 31. PMID 37268445
- [Derived] Kallionpaa RE, Valli K, Scheinin A, Langsjo J, Maksimow A, Vahlberg T, Revonsuo A, Scheinin H, Mashour GA, Li D. Alpha band frontal connectivity is a state-specific electroencephalographic correlate of unresponsiveness during exposure to dexmedetomidine and propofol. Br J Anaesth. 2020 Oct;125(4):518-528. doi: 10.1016/j.bja.2020.05.068. Epub 2020 Aug 7. PMID 32773216
- [Derived] Kallioinen M, Scheinin A, Maksimow M, Langsjo J, Kaisti K, Takala R, Vahlberg T, Valli K, Salmi M, Scheinin H, Maksimow A. The influence of dexmedetomidine and propofol on circulating cytokine levels in healthy subjects. BMC Anesthesiol. 2019 Dec 5;19(1):222. doi: 10.1186/s12871-019-0895-3. PMID 31805854
- [Derived] Kallionpaa RE, Scheinin A, Kallionpaa RA, Sandman N, Kallioinen M, Laitio R, Laitio T, Kaskinoro K, Kuusela T, Revonsuo A, Scheinin H, Valli K. Spoken words are processed during dexmedetomidine-induced unresponsiveness. Br J Anaesth. 2018 Jul;121(1):270-280. doi: 10.1016/j.bja.2018.04.032. Epub 2018 May 23. PMID 29935582
- [Derived] Radek L, Kallionpaa RE, Karvonen M, Scheinin A, Maksimow A, Langsjo J, Kaisti K, Vahlberg T, Revonsuo A, Scheinin H, Valli K. Dreaming and awareness during dexmedetomidine- and propofol-induced unresponsiveness. Br J Anaesth. 2018 Jul;121(1):260-269. doi: 10.1016/j.bja.2018.03.014. Epub 2018 May 10. PMID 29935581
- See also: Research Group Home Page — http://www.turkupetcentre.fi/index.php?option=com_content&view=article&id=268&Itemid=27